CLINICAL TRIAL: NCT01552330
Title: Open-Label Study to Evaluate Potential Pharmacokinetic Interaction of Orally Administered Primaquine and Pyronaridine-Artesunate in Healthy Adult Subjects
Brief Title: Pharmacokinetic Study of Primaquine and Pyronaridine-Artesunate in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP-C-016-11
Record Dates: First submitted 2012-03-01; First posted 2012-03-13 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Primaquine; Pyronaridine-artesunate
MeSH Terms: interventions — Primaquine; pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Primaquine only followed by Pyronaridine-Artesunate and followed by Primaquine together with Pyronaridine-Artesunate.
  Interventions: Drug: Primaquine and Pyronaridine-artesunate
- Group B (Active Comparator): Primaquine only followed by Primaquine together Pyronaridine-Artesunate and followed by Pyronaridine-Artesunate only.
  Interventions: Drug: Primaquine and Pyronaridine-Artesunate

INTERVENTIONS:
Drug: Primaquine and Pyronaridine-artesunate — Subject will receive primaquine (PQ) then receive pyronaridine-artesunate (PA)after 1 week washout period and receive PQ together with PA for the third regimen after 8 weeks washout period
  Primaquine:
  - Dosage: 2 tablets
  and
  Pyronaridine-Artesunate:
  - Dosage: 3 tablets
  Other Names: Pyramax
  Arms: Group A
Drug: Primaquine and Pyronaridine-Artesunate — Subject will receive primaquine (PQ) then receive PQ together dihydroartemisinin-piperaquine (DHA-PQP) after 1 week washout period and receive DHA-PQP for the third regimen after 8 weeks washout period.
  Primaquine:
  - Dosage: 2 tablets
  and
  Pyronaridine-Artesunate:
  - Dosage: 3 tablets
  Other Names: Pyramax
  Arms: Group B

SUMMARY:
The observed changes of P. falciparum sensitivity to artemisinin lead to the intensification of early detection as well as treatment monitoring in malaria infection. It is widely accepted that the development of resistance can be delayed by the use of combination therapy, especially combinations that include artemisinin derivatives (acts). As the resistance problem is considered extremely serious; as a consequence, who has recommended that all monotherapy for malaria should be stopped.

Current WHO guidelines recommend that the drug combination regimens using ACT with effective partner medicines should be used to decrease the risk of development or spreading of artemisinin resistance.

DETAILED DESCRIPTION:
Current WHO guidelines recommend that the drug combination regimens using ACT with effective partner medicines should be used to decrease the risk of development or spreading of artemisinin resistance.

Pyronaridine (PP) and artesunate (AS) are antimalarial agents with a history of clinical use both separately and in combination with other drugs. Each drug has powerful anti-schizonticidal actions. The action of artesunate is a rapid knock-down of the parasites, after which the drug is rapidly cleared as it has a short systemic half-life. Pyronaridine is also effective in the short-term but has an intermediate blood half-life thus providing a sustained schizonticidal effect. The aim of the fixed dose combination of pyronaridine and artesunate (PA or PYRAMAX®) in the treatment of uncomplicated acute malaria is to provide a rapid reduction in parasitemia with a short-term regimen, thereby improving compliance and reducing the risk of recrudescence through the slower elimination of pyronaridine. Doses have been selected to be in line with current prescribing practice for these agents when used as mono-therapy.

Primaquine (PQ) is an effective gametocytocide for P. falciparum transmission prevention and as tissue killing for the radical cure in P. vivax and P. ovale infection. It will be given only in the presence of other antimalarials, so it is necessary to study the drug interactions between primaquine, pyronaridine and artesunate. It is inevitable that in the near future, pyronaridine-artesunate (PA) and primaquine (PQ) combination treatment will become necessary. These drugs are metabolized by cytochrome P450 enzymes which potentially causes pharmacokinetic alteration and clinically significant drug-drug interactions that can lead to unanticipated adverse reactions or therapeutic failures because of the suboptimal exposure of the parasite.

This study is planned to evaluate potential pharmacokinetic interaction of orally administered primaquine and pyronaridine-artesunate (PYRAMAX®) in healthy adult subjects. The results of these interaction studies are important in order to provide clinical guidance for the optimum combination primaquine and pyronaridine-artesunate (PYRAMAX®) treatment regimens in malaria infections.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination.
2. Males and Females aged between 18 years to 60 years.
3. Males and Females weighing between 45-64 kilograms.
4. A female is eligible to enter and participate in this study if she is:

   * of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy
   * or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
   * or of childbearing potential, has a negative serum pregnancy test at screening and prior to start the study drug in each period, and abstain from sexual intercourse or agrees to using effective contraceptive methods (e.g., intrauterine device, hormonal contraceptive drug, tubal ligation or female barrier method with spermicide) during the study until completion of the follow-up procedures
5. A male is eligible to enter and participate in this study if he: agrees to abstain from (or use a condom during) sexual intercourse with females of childbearing potential or lactating females; or is willing to use a condom/spermicide, during the study until completion of the follow-up procedures.
6. Provide a signed and dated written informed consent prior to study participation.
7. Normal electrocardiogram (ECG) with QTc <450 msec.
8. Willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. The subject has evidence of active substance abuse that may compromise safety, pharmacokinetics, or ability to adhere with protocol instructions.
3. A positive pre-study hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
4. Subjects with a personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de pointes (heart failure, hypokalemia) or with a family history of sudden cardiac death.
5. A creatinine clearance <70 mL/min as determined by Cockcroft-Gault equation:

   CLcr (mL/min) = (140 - age) * Wt / (72 * Scr) (multiply answer by 0.85 for females) Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dL [Cockcroft, 1976].
6. History of alcohol or substance abuse or dependence within 6 months of the study.
7. Use of prescription or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety; the investigator will take advice from the manufacturer representative as necessary.
8. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
9. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample during each regimen.
10. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period. Note: This does not include plasma donation.
11. Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
12. Lack of suitability for participation in this study, including but not limited to, unstable medical conditions, systemic disease manifested by tendency to granulocytopenia e.g. rheumatoid arthritis and lupus erythematosus that in the opinion of the investigator would compromise their participation in the trial.
13. AST or ALT > 1 x upper limit of normal (ULN).
14. Subjects with history of renal disease, hepatic disease, and/or cholecystectomy
15. G6PD deficient detected by Beutler's dye test.
16. Abnormal methemoglobin level.
17. History of antimalarial drugs use including but not limited to mefloquine, chloroquine, primaquine, artesunate, piperaquine and pyronaridine treatment within 12 months.
18. Subject who received quinacrine in last 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Area under curve for Primaquine | 42 days
  Area under the concentration-time curve (AUC) for primaquine when given alone or together with Pyronaridine-Artesunate.
Area under cure for Pyronaridine-Artesunate | 42 days
  Area under the concentration-time curve (AUC) for pyronaridine when given alone as Pyronaridine-Artesunate (PA) or together with primaquine.

SECONDARY OUTCOMES:
Area under curve for Artesunate | 42 days
  Area under the concentration-time curve (AUC) for Artesunate/DHA when given alone as Pyronaridine-Artesunate or together with primaquine.
Maximum concentration and Area under curve for Primaquine and its metabolites | 42 days
  Primaquine enantiomers and Pyronaridine Cmax; carboxyprimaquine (and other detectable major metabolites) Cmax, AUC.
Assesment of safe and tolerability of Pyronaridine-Artesunate | 42 days
  Collecting number of adverse events, clinical laboratory, and vital signs assessments, ECG.
Pharmacogenetic polymorphisms | 42 days
  Pharmacogenetic polymorphisms in the case of unusually high or low drug levels.

CONTACTS AND LOCATIONS:
Overall Officials: Podjanee Jittamala, MD, Principal Investigator — Mahidol University
Locations (1):
- Hospital of Tropical Diseases, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Derived] Jittamala P, Pukrittayakamee S, Ashley EA, Nosten F, Hanboonkunupakarn B, Lee SJ, Thana P, Chairat K, Blessborn D, Panapipat S, White NJ, Day NP, Tarning J. Pharmacokinetic interactions between primaquine and pyronaridine-artesunate in healthy adult Thai subjects. Antimicrob Agents Chemother. 2015 Jan;59(1):505-13. doi: 10.1128/AAC.03829-14. Epub 2014 Nov 10. PMID 25385096